CLINICAL TRIAL: NCT00636454
Title: Coping Skills Training for Arthritis: An Effectiveness Trial
Brief Title: Effectiveness of a Training Program in Improving Coping Skills in People With Arthritis Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Joan Broderick, Principal Investigator, National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AR054626 (NIH); R01AR054626 (NIH); 1R01AR054626-01A1 (NIH); 3R01AR054626-03S2 (NIH)
Record Dates: First submitted 2008-03-12; First posted 2008-03-14 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Osteoarthritis
Keywords: OA; Pain; Cognitive Therapy; Behavior Therapy; Knee OA; Hip OA
MeSH Terms: conditions — Osteoarthritis; Pain; Osteoarthritis, Hip | interventions — galactosylceramide sulfotransferase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): This group will serve as the control group and will receive only the care usually given to OA patients.
  Interventions: Other: Usual care
- 2 (Experimental): This group will take part in the 10-session treatment program that will teach patients cognitive and behavioral skills to cope with pain.
  Interventions: Behavioral: Coping skills training (CST) for chronic pain

INTERVENTIONS:
Behavioral: Coping skills training (CST) for chronic pain — Participants will attend 10 sessions lasting between 45 and 60 minutes each. Topics will include relaxation training, managing activity cycles, and changing thought patterns to reduce the negative effects of pain.
  Arms: 2
Other: Usual care — Participants will receive the care usually given to patients with knee or hip OA.
  Arms: 1

SUMMARY:
Osteoarthritis (OA) is the leading cause of disability in the United States. Studies have shown that training patients to cope with pain improves physical and social functioning, increases self-efficacy, and reduces psychological distress. However, this type of training is not available to the vast majority of OA patients. This study will determine the effectiveness of a training program for coping with pain that will be administered in community medical practices.

A THIRD ARM OF THE TRIAL WAS FUNDED 09/09. TREATED PATIENTS WILL BE RANDOMIZED TO (1)A 4-MONTH COMPUTER-DRIVEN TELEPHONE PROGRAM TO ENHANCE MAINTANENCE OF TREATMENT GAINS OR (2)USUAL CARE. THIS ARM WILL ONLY BE CONDUCTED AT THE STONY BROOK SITE.

DETAILED DESCRIPTION:
OA affects approximately 60 percent of people older than 65 and can cause significant pain and impairment in functioning. Biomedical treatments are limited in their ability to curb OA disease progression and to eliminate pain and functional impairment. Consequently, health-related quality of life is often significantly impaired in people with arthritis. In academic research settings, pain coping skills training (CST) for arthritis improves the negative physical and social effects of OA. However, CST is not available to the vast majority of OA patients. Proving that CST is equally successful in community medical settings might make it more available to patients receiving care in these settings. Nurses with training in patient education are likely to be well-suited to deliver CST. This study will determine the effectiveness of CST for reducing arthritis pain when it is administered by nurse practitioners and registered nurses in community medical settings.

Participants in this study will be randomly assigned to either take part in a 10-session CST program for chronic pain or receive usual care. Participants in the treatment program will attend sessions in their doctor's offices. A nurse practitioner or registered nurse will meet with each participant for approximately 45 minutes each week to teach methods for management of pain associated with OA. Some of the strategies will include relaxation training, managing activity cycles, and changing thought patterns to reduce the negative effects of pain. Some sessions may be conducted on the phone rather than in person. All sessions will be tape-recorded for quality assurance purposes. Participants will be asked to practice coping skills between visits. At the end of the last visit, participants will spend an additional 60 minutes completing a booklet of questions about their health, pain levels, and response to the treatment program. Participants assigned to the usual care group will continue to see their healthcare providers as they normally would. They will not meet with the nurse or receive the CST. Assessments of pain, physical and psychological disability, self-efficacy, pain coping skills, and quality of life will be conducted for all participants pre-treatment, post-treatment, and at 6-month and 1-year follow-ups.

THE THIRD ARM OF THE TRIAL WILL PROVIDE 4 MONTHS OF PRE-RECORDED REVIEW OF COPING SKILLS TRAINING AS WELL AS DAILY RATINGS OF ARTHRITIS-RELATED PATIENT REPORTED OUTCOMES VIA A COMPUTER-DRIVEN TELEPHONE PROGRAM. PATIENTS ARE ASKED TO COMPLETE THE DAILY RATINGS AND CAN OPT TO LISTEN TO REVIEWS AND PRACTICE SESSIONS OF THE SKILLS THEY LEARNED WHILE RECEIVING CST TREATMENT FROM THE NURSE. AT THE END OF EACH MONTH, THE NURSE REVIEWS THE DAILY RATINGS AND PATIENT UTILIZATION OF THE REVIEW PROGRAM AND RECORDS A PERSONALIZED MESSAGE TO THE PATIENT TO IDENTIFY IMPORTANT PATTERNS AND TO ENCOURAGE USE OF THE PROGRAM.

TWO SETS OF PATIENTS WILL BE RANDOMIZED INTO THIS THIRD ARM OF THE TRIAL: THOSE WHO COMPLETED THE 12-MONTH STUDY ASSESSMENT ("OLD PATIENTS") AND THOSE WHO ARE JUST ENTERING THE TRIAL ("NEW PATIENTS"). THE FORMER WILL DETERMINE IF THE TELEPHONE MAINTANENCE PROGRAM IS EFFECTIVE FOR PATIENTS WHO COMPLETED CST TREATMENT OVER A YEAR AGO; THE LATTER WILL DETERMINE IF IT IS EFFECTIVE FOR PATIENTS WHEN USED IMMEDIATELY AT THE END OF CST TREATMENT. A TOTAL OF 50 PATIENTS WILL PARTICIPATE IN THE THIRD ARM OF THE TRIAL. OUTCOMES WILL BE MEASURED PRIOR TO THE START OF THE TELPHONE MAINTANENCE PROGRAM AND AT THE END OF THE 4-MONTH PROGRAM. OUTCOME ASSESSMENTS WILL BE IDENTICAL TO THOSE IN THE MAIN TRIAL.

ELIGIBILITY:
Inclusion Criteria:

* Patient in one of the two recruitment community clinics
* Diagnosis of knee or hip OA
* History of pain greater than or equal to a 4 on a 10-point scale for at least 6 months prior to study entry
* Able to read, write, and understand English
* Absence of significant psychiatric or cognitive dysfunction
* Able to attend 10 treatment sessions
* Access to telephone to complete interactive voice response (IVR) ratings and possible phone sessions
* Completion of baseline assessment

Exclusion Criteria:

* Scheduled for joint replacement surgery within the 18 months following study entry

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2008-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Pain | Measured pre-treatment, post-treatment, and at 6-month and 1-year follow-ups
Physical disability | Measured pre-treatment, post-treatment, and at 6-month and 1-year follow-ups
Psychological disability | Measured pre-treatment, post-treatment, and at 6-month and 1-year follow-ups
Self-efficacy | Measured pre-treatment, post-treatment, and at 6-month and 1-year follow-ups
Use of coping strategies | Measured pre-treatment, post-treatment, and at 6-month and 1-year follow-ups
Quality of life | Measured pre-treatment, post-treatment, and at 6-month and 1-year follow-ups

SECONDARY OUTCOMES:
Cost effectiveness of treatment | Measured at 12-month follow-up
RE-AIM measures of treatment fidelity | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Joan E. Broderick, PhD, Principal Investigator — Stony Brook University
Locations (3):
- United States (3):
  - Stony Brook Primary Care, Setauket, New York
  - Rheumatology Associates of Long Island, Smithtown and Port Jefferson, New York
  - Piedmont Primary Care, Danville, Virginia